CLINICAL TRIAL: NCT06392698
Title: Translation and Validation of the Dutch Surgical Fear Questionnaire in a Danish Population
Brief Title: The Danish Version of the Surgical Fear Questionnaire
Status: Completed | Type: Observational
Sponsor: Gødstrup Hospital (Other)
Collaborators: University of Aarhus (Other); Maastricht University Medical Center (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Brigitta Rasmussen Villumsen, Principal Investigator, Gødstrup Hospital
Other Study IDs: 1-16-02-82-24.
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Fear Anxiety; Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this translation and validation study is to make the The Dutch Surgical Fear Questionnaire (SFQ) applicable in adult Danish speaking patients referred to surgery.

After succesful translation of the SFQ, 200 adult patients referred to surgery at Gødstrup Hospital will be invited to answer the SFQ as well as two other questionnaires for the validation: The Pain Catastrophizing Scale (PCS) and The Hospital Anxiety and Depression Scale (HADS).

Statistical analysis will be performed to assess the correlation between the scales and thus the validity of the SFQ.

DETAILED DESCRIPTION:
Some of the instruments for assessing surgical fear are the Amsterdam Preoperative Anxiety and Information Scale (APAIS), the Hospital anxiety and depression scale (HADS), the State-Trait Anxiety Inventory (STAI) and the Visual Analog Scale assessing Anxiety (VAS-A). However, HADS, STAI and VAS-A ask questions not particular related to perioperative procedures and thus seem too generic and APAIS seems unspecific despite questions directly related to anaesthesia and the surgical procedure. The Dutch Surgical Fear Questionnaire (SFQ) was developed to be suitable for general use among all types of adult surgery patients to assess self-reported surgical fear, and to cover a broad range of short-term and long-term surgery-related fears.

The translation and validation follows the standardized multistep process outlined by Cha, Kim, and Erlen: 1) forward translation, 2) backward translation by native speakers, 3) a test of the translation in a pilot population of adults referred to surgery at Gødstrup Hospital, and 4) validation in a clinical population.

For the validation of quantitatively measured clinical variables (clinimetric validation), convergent validity will be assessed between SFQ, the Pain Catastrophizing Scale (PCS) and the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A). The Cronbach's alpha test will be employed to assess the internal consistency of the SFQ subscales and the overall score.

Approval of the study has been obtained from the Institutional Review Board at Central Denmark Region. Informed consent will be obtained from all participants prior to inclusion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to read and understand Danish
* Cognitive well-functioning
* No previously or ongoing diagnosed mental disorders
* Consent to participate in the study.

Exclusion Criteria:

* Any patient who in the opinion of the investigator does not comply with the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients referred to surgery at Gødstrup Hospital
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Correlations between the SFQ and the PCS and SFQ and the anxiety subscale of the HADS | 2025
  Assement will be conducted using Spearman correlation analysis
Internal consistency | 2025
  The Cronbach's alpha test will be employed to assess the internal consistency of the SFQ
Confirmatory factor analysis | 2025
  A confirmatory factor analysis (CFA) will be conducted to investigate whether the factor structure confirms the original Dutch version.
Cut-off values for item-specific clinically significant surgical fear | 2025
  For each of the 8 items on the Surgical Fear Questionnaire, a cut-off value between 0-10 will be calculated to determine clinically relevant surgical fear.

SECONDARY OUTCOMES:
Frequency distribution | 2025
  For each of the 8 items on the Surgical Fear Questionnaire minimum and maximum score, mean, median and Interquartile Range (IQR) will be calculated.
Floor and ceiling effect | 2025
  Number and percentages of respondents who score the lowest value (=0) and highest value (=10) on each individual item on the Surgical Fear Questionnaire
Fear of short-term consequences of surgery | 2025
  The first 4 items on the Surgical Fear Questionnaire constitue a subscale related to the fear of short-term consequences of surgery. Each item is rated on a numerical rating scale 0-10 where 0 is the lowest and 10 the highest level of fear. The score on the subscale ranges from 0-40.
  Minimum, maximun, meand, standard deviation, median and Interquartile Range will be calculated.
Fear of long-term consequences of surgery | 2025
  The last 4 items on the Surgical Fear Questionnaire constitute a subscale related to the fear of long-term consequences of surgery. Each item is rated on a numeric rating scale ranging from 0-10 where 0 is = not afraid and 10 = very afraid. The score on the subscale range from 0-40.
  Minimum, maximum, meand, standard deviation, median and Interquartile Range will be calculated.
Scores on the Surgical Fear Questionnaire | 2025
  The questionnaire contains 8 items and each item is rated on a numeric rating scale ranging from 0 (not afraid) to 10 (very afraid). The total score ranges from 0 to 80, where higher score means higher level of fear.
  Minimum, maximum, meand, standard deviation, median and Interquartile Range will be calculated.
Scores on the Pain Catastrophizing Scale (PCS) | 2025
  Pain Catastrophizing consists of three distinct, but interrelated concepts: rumination, magnification and helplessness which construct are assessed with three subscales on the 13-item Pain Catastrophizing Scale (PCS). Respondents provide answers on a 5-point Likert scales ranging from 0 (not at all) to 4 (all the time). Higher score indicate higher level of pain catastrophizing. The scale ranges from 0-52 Minimum, maximum, mean, standard deviation, median and Interquartile Range will be calculated.
Scores on the Hospital Depression and Anxiety Scale (HADS) | 2025
  The HADS is commonly used in non-psychiatric hospital settings to identify anxiety disorders and depression. It comprises two subscales, Anxiety and Depression, each consisting of 7 items. Respondents provide answers on a 4-point Likert scale ranging from 0 to 3. Separate scores are computed for the Anxiety and Depression subscales, with higher scores indicating greater symptom severity. The scores range from 0-21 on each subscale.
  Minimum, maximum, mean, standard deviation, median and Interquartile Range will be calculated
The association between surgical fear and gender | 2025
  The Kruskal-Wallis test will be applied to calculated the association.
The correlation between surgical fear and age | 2025
  The Spearman rank correlation will be applied to calculate the association.
The association between surgical fear and educational level | 2025
  The Kruskal-Wallis test will be applied to calculate the association.
The association between surgical fear and civil status | 2025
  The Kruskal-Wallis test will be applied to calculate the association.
The association between surgical fear and type of admission (day surgery versus hospitalised overnight) | 2025
  The Mann-Whitney U Test will be applied to calculate the association
The association between surgical fear and cancer versus non-cancer surgery | 2025
  The Kruskal-Wallis test will be applied to calculate the association
The association between surgical fear and previous surgery versus no previous surgery | 2025
  The Mann-Whitney U Test will be applied to calculate the association.
The association between surgical fear and type of anaesthesia | 2025
  Three groups of anaesthesia:
  1. General alone, vs
  2. General plus regional with or without sedation vs
  3. Regional or local with or without sedation The Kruskal-Wallis Test will be applied for the calculations. In case of significant results the test will be followed by Dunn's test with Bonferroni correction to determine which specific groups are different.
The association between surgical fear and postoperative pain | 2025
  A logistic regression analysis will be applied to calculate the likelihood of postoperative pain score based on preoperative surgical fear.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta R Villumsen, Postdoc, Principal Investigator — Gødstrup Hospital
Locations (1):
- Gødstrup Hospital, Herning, Denmark

REFERENCES:
- [Background] Theunissen M, Peters ML, Schouten EG, Fiddelers AA, Willemsen MG, Pinto PR, Gramke HF, Marcus MA. Validation of the surgical fear questionnaire in adult patients waiting for elective surgery. PLoS One. 2014 Jun 24;9(6):e100225. doi: 10.1371/journal.pone.0100225. eCollection 2014. PMID 24960025
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Pinto PR, McIntyre T, Almeida A, Araujo-Soares V. The mediating role of pain catastrophizing in the relationship between presurgical anxiety and acute postsurgical pain after hysterectomy. Pain. 2012 Jan;153(1):218-226. doi: 10.1016/j.pain.2011.10.020. Epub 2011 Nov 23. PMID 22115922
- [Background] Cha ES, Kim KH, Erlen JA. Translation of scales in cross-cultural research: issues and techniques. J Adv Nurs. 2007 May;58(4):386-95. doi: 10.1111/j.1365-2648.2007.04242.x. Epub 2007 Apr 17. PMID 17442038